CLINICAL TRIAL: NCT00577473
Title: A Double-blind, Randomized, 6 Week, Parallel-group Design Clinical Trial in Patients With Mildly to Moderately Active Ulcerative Colitis to Assess the Safety and Efficacy of Asacol 4.8 g/Day Versus Asacol 2.4 g/Day
Brief Title: Safety and Efficacy of Asacol 4.8 g/Day Versus Asacol 2.4 g/Day (ASCEND I)
Acronym: ASCEND I
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Warner Chilcott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2000083
Record Dates: First submitted 2007-12-19; First posted 2007-12-20 (Estimated); Results first posted 2011-06-22 (Estimated); Last update posted 2011-09-16 (Estimated); Status verified 2011-09

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Mesalamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): mesalamine 2.4 g/day (400 mg tablet) for 6 weeks
  Interventions: Drug: mesalamine
- 2 (Experimental): mesalamine 4.8 g/day (800 mg tablet) for 6 weeks
  Interventions: Drug: mesalamine

INTERVENTIONS:
Drug: mesalamine — mesalamine 2.4 g/day (400 mg tablet) for 6 weeks
  Arms: 1
Drug: mesalamine — mesalamine 4.8 g/day (800 mg tablet) for 6 weeks
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Asacol 4.8 g/day (800 mg tablet) versus Asacol 2.4 g/day (400 mg tablet

DETAILED DESCRIPTION:
This study is designed to evaluate the safety and efficacy of 4.8 g/day using 800 mg Asacol tablets as compared to 2.4g/day using 400 mg Asacol tablets in newly- and previously-diagnosed patients who are experiencing a flare-up of mildly to moderately active ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of ulcerative colitis

Exclusion Criteria:

* a history of allergy or hypersensitivity to salicylates or aminosalicylates;
* a history of extensive small bowel resection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2001-02; Primary Completion 2003-02 (Actual); Study Completion 2003-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery Kralstein, MD, Study Director — Procter and Gamble
Locations (44):
- United States (44):
  - Research Site, Birmingham, Alabama
  - Research Site, Anaheim, California
  - Research Site, Sacramento, California
  - Research Site, San Francisco, California
  - Research Site, Denver, Colorado
  - Research Facility, Golden, Colorado
  - Research Site, Bridgeport, Connecticut
  - Research Site, Fort Myers, Florida
  - Research Site, Hollywood, Florida
  - Research Site, Jupiter, Florida
  - Research Site, Miami, Florida
  - Research Facility, Atlanta, Georgia
  - Research Facility, Decatur, Georgia
  - Research Site, Arlington Heights, Illinois
  - Research Site, Moline, Illinois
  - Research Site, Rockford, Illinois
  - Research Site, Wichita, Kansas
  - Research Site, Metairie, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, Laurel, Maryland
  - Research Site, Detroit, Michigan
  - Research Site, New Brunswick, New Jersey
  - Research Site, Somerville, New Jersey
  - Research Site, Great Neck, New York
  - Research Site, Pomona, New York
  - Research Facility, Poughkeepsie, New York
  - Research Site, Raleigh, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Tulsa, Oklahoma
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Facility, Memphis, Tennessee
  - Research Facility, Nashville, Tennessee
  - Research Site, Fort Worth, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Burlington, Vermont
  - Research Site, Charlottesville, Virginia
  - Research Facility, Falls Church, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Tacoma, Washington
  - Research Site, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Orchard TR, van der Geest SA, Travis SP. Randomised clinical trial: early assessment after 2 weeks of high-dose mesalazine for moderately active ulcerative colitis - new light on a familiar question. Aliment Pharmacol Ther. 2011 May;33(9):1028-35. doi: 10.1111/j.1365-2036.2011.04620.x. Epub 2011 Mar 8. PMID 21385195
- [Derived] Lichtenstein GR, Ramsey D, Rubin DT. Randomised clinical trial: delayed-release oral mesalazine 4.8 g/day vs. 2.4 g/day in endoscopic mucosal healing--ASCEND I and II combined analysis. Aliment Pharmacol Ther. 2011 Mar;33(6):672-8. doi: 10.1111/j.1365-2036.2010.04575.x. Epub 2011 Jan 23. PMID 21255059

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Screening began 9 Feb 2001
Groups:
- Asacol 2.4 g/Day: 2 - 400 mg Asacol tablets and 2 placebo tablets (matching 800 mg Asacol tablet) 3 times daily for 6 weeks
- Asacol 4.8 g/Day: 2 - 800 mg Asacol tablets and 2 placebo tablets (matching 400 mg tablet) 3 times daily for 6 weeks
Period: Overall Study
Arm/Group | Asacol 2.4 g/Day | Asacol 4.8 g/Day
Started | 154 | 147
ITT Population | 150 | 136
Completed | 133 | 123
Not Completed | 21 | 24
Not completed — Protocol Violation | 1 | 4
Not completed — Adverse Event | 8 | 5
Not completed — Withdrawal by Subject | 2 | 6
Not completed — Physician Decision | 2 | 2
Not completed — Lack of Efficacy | 8 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Asacol 2.4 g/Day | Asacol 4.8 g/Day | Total
Number analyzed (Participants) | 154 | 147 | 301
Age, Customized [Number; unit: Participants]
  18 - 64 years | 141 | 133 | 274
  >= 65 years | 13 | 14 | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 67 | 146
  Male | 75 | 80 | 155
Race/Ethnicity, Customized [Number; unit: Partcipants]
  Caucasian | 122 | 116 | 238
  Black or African American | 18 | 18 | 36
  Asian (Indian) | 2 | 2 | 4
  Asian (Oriental) | 1 | 0 | 1
  Hispanic | 10 | 9 | 19
  Multi-racial/other | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Classified as Treatment Success at Week 6, ITT Population
Description: Treatment Success - complete or partial response; Complete = complete resolution of clinical assessments (stool frequency, rectal bleeding, PFA [patient's functional assessment], sigmoidoscopy) and PGA (physician global assessment) = 0, Partial = improvement from baseline PGA score and improvement in at least 1 of the clinical assessments [decrease of at least 1 on scale] and no worsening [no score increases] of remaining clinical assessments. Each clinical assessment graded using scale 0/normal, better thru 3/severe, worse.
Time Frame: 6 weeks
Population: ITT Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Asacol 2.4 g/Day | Asacol 4.8 g/Day
Number analyzed (Participants) | 150 | 136
Percentage of Participants | 51.3 | 55.9
Statistical Analysis 1: Comparison: Asacol 2.4 g/Day vs Asacol 4.8 g/Day; It was assumed that the true rate of improvement for the 2.4 g/day treatment group is 40% and for the 4.8 g/day group is 60%. To detect a true difference of 20% between these 2 groups with a 2-sided test, type I error of 0.05 (α = 0.05), and power of 90%, 140 patients were required per group to complete the study. To account for a 10% dropout/withdrawal rate, approximately 308 patients were to be enrolled in the study; Test type: Superiority or Other; p = 0.4411, Chi-squared — 4.8 g/day compared to 2.4 g/day; Risk Difference (RD) = 0.0455, 95% CI 2-sided [-7.01 to 16.11]

2. Secondary Outcome: Percentage of Patients Classified as Treatment Success at Week 3, ITT Population
Description: as for outcome 1
Time Frame: 3 weeks
Population: ITT Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Asacol 2.4 g/Day | Asacol 4.8 g/Day
Number analyzed (Participants) | 150 | 137
Percentage of Participants | 42.0 | 38.7
Statistical Analysis 1: Comparison: Asacol 2.4 g/Day vs Asacol 4.8 g/Day; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5677, Chi-squared; Risk Difference (RD) = -0.0331, 95% CI 2-sided [-14.67 to 8.04]

3. Secondary Outcome: Physician's Global Assessment (PGA) Percentage of Patients Improved at Week 3, All Randomized Patients
Description: PGA - 0-quiescent disease activity (all 0's) , 1-mild (mostly 1's), 2-moderate (mostly 2's), 3-severe (mostly 3's) based upon on scoring for stool frequency, rectal bleeding, PFR (patient's functional assessment - 0-well, 1-fair, 2-poor, 3-terrible), sigmoidoscopy findings. Improvement defined as either complete response (remission, score = 0) or partial response (improvement on treatment). Scoring Scale: 0-good thru 3-worse.
Time Frame: Week 3
Population: All Randomized Patients
Measure: Number; unit: Percentage of Participants
Arm/Group | Asacol 2.4 g/Day | Asacol 4.8 g/Day
Number analyzed (Participants) | 154 | 147
Percentage of Participants | 49.3 | 44.8
Statistical Analysis 1: Comparison: Asacol 2.4 g/Day vs Asacol 4.8 g/Day; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4730, Chi-squared; Risk Difference (RD) = -0.0445, 95% CI 2-sided [-16.6 to 7.7]

4. Secondary Outcome: Physician's Global Assessment (PGA) Percentage of Patients Improved at Week 6, All Randomized Patients
Description: PGA - 0-quiescent disease activity (all 0's) , 1-mild (mostly 1's), 2-moderate (mostly 2's), 3-severe (mostly 3's) based upon on scoring for stool frequency, rectal bleeding, PFR (patient's functional assessment - 0-well, 1-fair, 2-poor, 3-terrible), sigmoidoscopy findings. Improvement defined as complete response (remission, score = 0) or partial response (improvement on treatment). Scoring Scale: 0-good thru 3-worse.
Time Frame: Week 6
Population: All Randomized Patients
Measure: Number; unit: Percentage of Participants
Arm/Group | Asacol 2.4 g/Day | Asacol 4.8 g/Day
Number analyzed (Participants) | 154 | 147
Percentage of Participants | 61.4 | 64.8
Statistical Analysis 1: Comparison: Asacol 2.4 g/Day vs Asacol 4.8 g/Day; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5761, Chi-squared; Risk Difference (RD) = 0.0339, 95% CI 2-sided [-8.48 to 15.26]

5. Secondary Outcome: Stool Frequency Improvement at Week 3, All Randomized Patients (Percentage)
Description: 0: normal stool frequency per day, 1: 1-2 stools greater than normal per day, 2: 3-4 stools greater than normal per day, 3: 5 or more stools greater than normal per day, Scoring Scale: 0-good thru 3-worse.
Time Frame: Week 3
Population: All Randomized Patients
Measure: Number; unit: Percentage of Participants
Arm/Group | Asacol 2.4 g/Day | Asacol 4.8 g/Day
Number analyzed (Participants) | 154 | 147
Percentage of Participants | 46.7 | 54.3
Statistical Analysis 1: Comparison: Asacol 2.4 g/Day vs Asacol 4.8 g/Day; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2150, Chi-squared; Risk Difference (RD) = 0.0766, 95% CI 2-sided [-4.41 to 19.74]

6. Secondary Outcome: Stool Frequency Improvement at Week 6, All Randomized Patients (Percentage)
Description: as for outcome 5
Time Frame: Week 6
Population: All Randomized Patients
Measure: Number; unit: Percentage of Participants
Arm/Group | Asacol 2.4 g/Day | Asacol 4.8 g/Day
Number analyzed (Participants) | 154 | 147
Percentage of Participants | 63.2 | 66.7
Statistical Analysis 1: Comparison: Asacol 2.4 g/Day vs Asacol 4.8 g/Day; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5569, Chi-squared; Risk Difference (RD) = 0.0351, 95% CI 2-sided [-8.18 to 15.20]

7. Secondary Outcome: Rectal Bleeding Improvement at Week 3, All Randomized Patients (Percentage)
Description: 0: no blood seen, 1: streaks of blood with stool less than half of the time, 2: obvious blood with stool most of the time, 3: blood alone passed, Scoring Scale: 0-good thru 3-worse.
Time Frame: Week 3
Population: All Randomized Patients
Measure: Number; unit: Percentage of Participants
Arm/Group | Asacol 2.4 g/Day | Asacol 4.8 g/Day
Number analyzed (Participants) | 154 | 147
Percentage of Participants | 48.1 | 59.1
Statistical Analysis 1: Comparison: Asacol 2.4 g/Day vs Asacol 4.8 g/Day; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0769, Chi-squared; Risk Difference (RD) = 0.1091, 95% CI 2-sided [-1.10 to 22.91]

8. Secondary Outcome: Rectal Bleeding Improvement at Week 6, All Randomized Patients (Percentage)
Description: 0-no blood seen, 1- streaks of blood with stool less than half of the time, 2- obvious blood with stool most of the time, 3- blood alone passed. Scoring Scale: 0-good thru 3-worse.
Time Frame: Week 6
Population: All Randomized Patients
Measure: Number; unit: Percentage of Participants
Arm/Group | Asacol 2.4 g/Day | Asacol 4.8 g/Day
Number analyzed (Participants) | 154 | 147
Percentage of Participants | 60.2 | 71.5
Statistical Analysis 1: Comparison: Asacol 2.4 g/Day vs Asacol 4.8 g/Day; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0551, Chi-squared; Risk Difference (RD) = 0.1139, 95% CI 2-sided [-0.13 to 22.92]

9. Secondary Outcome: Improvement in Patient's Functional Assessment (PFA) at Week 3, All Randomized Patients (Percentage)
Description: 0-generally well, 1-fair, 2-poor, 3-terrible
Time Frame: Week 3
Population: All Randomized Patients
Measure: Number; unit: Percentage of Participants
Arm/Group | Asacol 2.4 g/Day | Asacol 4.8 g/Day
Number analyzed (Participants) | 154 | 147
Percentage of Participants | 42.2 | 49.6
Statistical Analysis 1: Comparison: Asacol 2.4 g/Day vs Asacol 4.8 g/Day; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2306, Chi-squared; Risk Difference (RD) = 0.0738, 95% CI 2-sided [-4.66 to 19.43]

10. Secondary Outcome: Improvement in Patient's Functional Assessment (PFA) at Week 6, All Randomized Patients (Percentage)
Description: 0-generally well, 1-fair, 2-poor, 3-terrible
Time Frame: Week 6
Population: All Randomized Patients
Measure: Number; unit: Percentage of Participants
Arm/Group | Asacol 2.4 g/Day | Asacol 4.8 g/Day
Number analyzed (Participants) | 154 | 147
Percentage of Participants | 54.1 | 60.7
Statistical Analysis 1: Comparison: Asacol 2.4 g/Day vs Asacol 4.8 g/Day; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2931, Chi-squared; Risk Difference (RD) = 0.0652, 95% CI 2-sided [-5.60 to 18.64]

11. Secondary Outcome: Improvement in Patient's Sigmoidoscopy Assessment Score at Week 3, All Randomized Patients (Percentage)
Description: 0-normal (intact vascular pattern, no friability or granularity), 1-mild (erythema; diminished or absent vascular markings; mild granularity; friability), 2-moderate (marked erythema, granularity; absent vascular markings; bleeds with minimal trauma; no ulcerations), 3-severe (spontaneous bleeding, ulcerations). Scoring Scale: 0-good thru 3-worse.
Time Frame: Week 3
Population: All Randomized Patients
Measure: Number; unit: Percentage of Participants
Arm/Group | Asacol 2.4 g/Day | Asacol 4.8 g/Day
Number analyzed (Participants) | 154 | 147
Percentage of Participants | 51.5 | 52.0
Statistical Analysis 1: Comparison: Asacol 2.4 g/Day vs Asacol 4.8 g/Day; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9349, Chi-squared; Risk Difference (RD) = 0.0051, 95% CI 2-sided [-11.67 to 12.69]

12. Secondary Outcome: Improvement in Patient's Sigmoidoscopy Assessment Score at Week 6, All Randomized Patients (Percentage)
Description: as for outcome 11
Time Frame: Week 6
Population: All Randomized Patients
Measure: Number; unit: Percentage of Participants
Arm/Group | Asacol 2.4 g/Day | Asacol 4.8 g/Day
Number analyzed (Participants) | 154 | 147
Percentage of Participants | 66.7 | 73.2
Statistical Analysis 1: Comparison: Asacol 2.4 g/Day vs Asacol 4.8 g/Day; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2583, Chi-squared; Risk Difference (RD) = 0.0650, 95% CI 2-sided [-4.72 to 17.73]

ADVERSE EVENTS:
Time Frame: 6 week treatment period
Description: Screening started February 2001, study completed November 2002
Arm/Group | Asacol 2.4 g/Day | Asacol 4.8 g/Day
Serious Adverse Events (participants affected / at risk) | 3/154 | 1/147
Other Adverse Events (participants affected / at risk) | 56/154 | 48/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Asacol 2.4 g/Day (N=154) | Asacol 4.8 g/Day (N=147)
Uterine Fibroids Exacerbation (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian Cyst Exacerbation (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Worsening of Ulcerative Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal Bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal Pain, Left Side (Vascular disorders) | 1 (1) | 0 (0)
Cholecystitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain, Right Upper Quadrant (Nervous system disorders) | 1 (1) | 0 (0)
Epigastric Pain (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Asacol 2.4 g/Day (N=154) | Asacol 4.8 g/Day (N=147)
Headache (Nervous system disorders) | 9 | 8
Nausea (Gastrointestinal disorders) | 2 | 9
Abdominal Pain (Gastrointestinal disorders) | 7 | 4
Infection (Infections and infestations) | 5 | 5
Diarrhea (Gastrointestinal disorders) | 5 | 4
Flatulence (Gastrointestinal disorders) | 3 | 6
Colitis Ulcer (Gastrointestinal disorders) | 6 | 2
Vomiting (Gastrointestinal disorders) | 1 | 6
Rash (Skin and subcutaneous tissue disorders) | 3 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Dizziness (Nervous system disorders) | 4 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 3
Flu Syndrome (Infections and infestations) | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less